CLINICAL TRIAL: NCT02461056
Title: Synergistic Effect of Ibuprofen and Hydromorphone for Postoperative Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Hyun Joo Ahn, Assoicate professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2014-03-108
Record Dates: First submitted 2015-05-28; First posted 2015-06-03 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-05

CONDITIONS: Breast Cancer
Keywords: ibuprofen; hydromorphone; drug interactions
MeSH Terms: conditions — Breast Neoplasms | interventions — Ibuprofen; Hydromorphone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ibuprofen (Active Comparator): Ibuprofen: Patients receive ibuprofen 50 mg, 100 mg, 200 mg, 400mg or 800 mg intravenously once at post-anesthesia care unit.
  Interventions: Drug: Ibuprofen
- hydromorphone (Active Comparator): Hydromorphone: Patients receive hydromorphone 0.25 mg, 0.5 mg, 1 mg, 1.5 mg, or 2 mg intravenously once at post-anesthesia care unit.
  Interventions: Drug: Hydromorphone
- ibuprofen+hydromorphone (Active Comparator): Ibuprofen+Hydromorphone: Patients receive ibuprofen 25 mg + hydromorphone 0.125 mg, ibuprofen 50 mg + hydromorphone 0.25 mg, ibuprofen 100 mg + hydromorphone 0.5 mg, ibuprofen 200 mg + hydromorphone 0.75 mg, or ibuprofen 400 mg + hydromorphone 1 mg intravenously once at post-anesthesia care unit.
  Interventions: Drug: Ibuprofen; Drug: Hydromorphone

INTERVENTIONS:
Drug: Ibuprofen — Drug was administered by the Dixon and Mood up-and-down method. Starting doses was ibuprofen 50 mg. The maximum doses was ibuprofen 800 mg. Combination index (CI) (additive: 0.9-1.1, synergism: <0.9, antagonism: >1.1), dose reduction index (DRI, a measure of how much the dose of each drug in a combination can be reduced), and isobologram were used to define the nature of their interaction.
  Other Names: Caldolor
  Arms: Ibuprofen; ibuprofen+hydromorphone
Drug: Hydromorphone — Drug was administered by the Dixon and Mood up-and-down method. Starting doses was hydromorphone 0.25 mg. The maximum doses was hydromorphone 2 mg. Combination index (CI) (additive: 0.9-1.1, synergism: <0.9, antagonism: >1.1), dose reduction index (DRI, a measure of how much the dose of each drug in a combination can be reduced), and isobologram were used to define the nature of their interaction.
  Other Names: Dilid
  Arms: hydromorphone; ibuprofen+hydromorphone

SUMMARY:
Intravenous form of ibuprofen is recently approved by FDA and reports are rare on the co-administration with opioids. The investigators searched whether intravenous ibuprofen-hydromorphone combination is synergistic, additive, or infra-additive on postoperative pain using combination index (CI), dose reduction index (DRI) and isobologram.

DETAILED DESCRIPTION:
Ninety patients, undergoing breast surgery, were included in one of the three groups (Ibuprofen, Hydromorphone, Ibuprofen+Hydromorphone groups). Positive analgesic efficacy was defined as a numeric rating scale (NRS) ≤3 on a 0-10 NRS, 30 min after the drug administration. Drug was administered by the Dixon and Mood up-and-down method. Starting doses were ibuprofen 50 mg, hydromorphone 0.25 mg, or ibuprofen 25 mg + hydromorphone 0.125 mg. The maximum doses were ibuprofen 800 mg, hydromorphone 2 mg, or ibuprofen 400 mg + hydromorphone 1 mg. Combination index (CI) (additive: 0.9-1.1, synergism: <0.9, antagonism: >1.1), dose reduction index (DRI, a measure of how much the dose of each drug in a combination can be reduced), and isobologram were used to define the nature of their interaction.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status І or ІІ who were able to communicate and understand the pain scales

Exclusion Criteria:

* any contraindication to the use of ibuprofen or hydromorphone
* a history of allergy or hypersensitivity
* a calculated creatinine clearance of <75 mL/min
* the presence or history of asthma, bleeding tendency, coronary artery bypass graft (CABG) surgery, heart failure, peptic ulcer disease, inflammatory bowel disease or any other gastrointestinal disorder, and renal or hepatic disease
* pregnancy
* age younger than 18 yr
* intraoperative use of regional anesthesia
* intraoperative administration of analgesics other than remifentanil
* postoperative pain ≤3 on a NRS in the post-anesthesia care unit (PACU)

Ages: 19 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2014-06; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Pain scores on the numeric rating scale (NRS) | postoperative 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Hyun Joo Ahn, Ph.D., Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung medical center, Seoul, South Korea